CLINICAL TRIAL: NCT06689592
Title: Untersuchung Der Durchführbarkeit Von TMS-Behandlungen Zuhause - Mobile Transkranielle Magnetstimulation "MTMS"
Brief Title: Mobile Transcranial Magnetic Stimulation
Acronym: MTMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Regensburg (Other)
Responsible Party: Principal Investigator, Berthold Langguth, MD, Ph.D., Clinical Professor, MD, Ph.D., University of Regensburg
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24-3652-101
Record Dates: First submitted 2024-11-12; First posted 2024-11-14 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mobile Transcranial Magnetic Stimulation (Experimental): Transcranial Magnetic Stimulation at home. Half of the SAINT protocol (Cole et al., 2020, 2022) is to be carried out. For this purpose, all 5 test subjects are treated with 5 sessions per day on 5 consecutive days (25 stimulations in total). An iTBS protocol (3 pulses at 50 Hz in 2 seconds, 8 seconds pause) with 1800 pulses (total duration: 10 minutes) should be used every hour with a break of 50 minutes (total of 9,000 pulses can be applied per day).
  Interventions: Device: Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation — Intermittent theta burst stimulation

SUMMARY:
For this study 5 patients will be treated with transcranial magnetic stimulation in their residence (home, nursing home).

DETAILED DESCRIPTION:
An investigation of the feasibility of rTMS treatments outside a clinical-medical context (e.g. in a residential facility and/or at the patient's home) is to be carried out (5 patients in total). Before the actual start of the study, the test subjects are informed in detail about the experimental setup and the methods used, as well as about contraindications and possible side effects. Following the information session, the test subjects sign a declaration of consent and complete questionnaires with relevant information (demographic data, health data to rule out serious illnesses and diagnostic questionnaires). On this day, a TMS test with a few test pulses is also planned in order to familiarize the test subjects with the TMS and to evaluate their tolerance. The stimulation intensity (so-called motor threshold) is also determined as part of this. In the following week, the TMS treatment is carried out on 5 consecutive days with a further visit. Following the preparations, a protocol modified from the Stanford Accelerated Intelligent Neuromodulation Therapy (SAINT) protocol is carried out. For this purpose, the test subjects are treated in 5 sessions per day on 5 consecutive days (25 stimulations in total). An iTBS protocol (3 bursts at 50 Hz in 2 seconds, 8 second pause) with 1800 pulses should be used every hour, which means that the duration of a stimulation is approximately 10 minutes and a total of 9,000 pulses could be applied per day.

The individual sessions are monitored by a Medbo Regensburg employee on site. There should be a break of 50 minutes between each hourly stimulation. After the treatment, a follow-up should take place after 4 weeks with questionnaires and a short verbal evaluation. Each subject can voluntarily terminate participation in the study at any time without giving reasons and without negative consequences (except for the lack of treatment). If the participant's compliance is severely impaired, the study may be terminated by the investigator.

ELIGIBILITY:
Inclusion Criteria:

* leading diagnosis of a depressive episode according to ICD-10 in the context of a uni- or bipolar disorder
* moderate depression according to the Hamilton Depression Rating Scale
* adult persons aged 18-80 of all genders
* place of residence in Germany and understanding of the German language sufficient to understand the information
* written declaration of consent

Exclusion Criteria:

* Fulfillment of the contraindications for TMS (electrical implants or metallic objects in the body such as pacemakers or insulin pumps, skin diseases on the head)
* The presence of a serious neurological disease (e.g. cerebrovascular events, neurodegenerative diseases, epilepsy, brain malformation, severe head injuries in the medical history)
* Participation in another study during the treatment
* Pregnancy and breastfeeding period

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2024-08-15 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Usability for the patients | 1 week
  Rating of the usability of the treatment with the user experience questionnaire [1-7, 26 items, the higher the better] and open feedback
Usability for the handlers/clinicians | 1 week
  Rating of the usability of the treatment (home treatment) with the user experience questionnaire [1-7, 26 items, the higher the better] and open feedback
Efficiancy 1 | 1 week
  Number of responders according the the clinical global impression change score for patients in the per protocol analysis
Efficiancy 2 | 1 week
  Effect size for change of depressivity for patients in the per protocol analysis measured with the Hamilton depression rating scale (21 items)
Stability of effects 1 | 5 weeks
  Number of responders according the the clinical global impression change score
Stability of effects 2 | 5 weeks
  Effect size for change of depressivity for patients in the per protocol analysis measured with the Hamilton depression rating scale (21 items)

SECONDARY OUTCOMES:
Course of the scores of the Hamilton depression rating scale | 1 week
  Depression rating scale (0-65, the lower the better)
Course of the scores of the Major Depression Inventory | 1 week
  Depression inventory (0-50, the lower the better)
Course of the scores of the WHO Quality of life scale (abbreviated Version) (WHOQOL-BREF) | 1 week
  Quality of life scale inventory (4-20, the higher the better)
Course of the scores of the Clincial Global Impression change | 1 week
  Clincial Global Impression (1-7, the lower the better)

CONTACTS AND LOCATIONS:
Overall Officials: Berthold Langguth, PhD, Principal Investigator — University of Regensburg
Locations (1):
- Department of Psychiatry and Psychotherapy, University of Regensburg, Regensburg, Germany, Regensburg, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No